CLINICAL TRIAL: NCT04285736
Title: The Efficacy of Oral Ivabradine in Patients Presenting With Acute Non ST-segment Elevation Myocardial Infarction (NSTEMI): Interventional Randomized Parallel Study
Brief Title: Efficacy of Oral Ivabradine in Patients Presenting With NSTEMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, Samar Farghali Farid, Professor and Head of Clinical Pharmacy Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL1200
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: NSTEMI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Ivabradine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Ivabradine Group (Experimental)
  Interventions: Drug: Ivabradine
- Group B Control Group (Active Comparator)
  Interventions: Drug: Ivabradine; Drug: Conventional Treatment

INTERVENTIONS:
Drug: Ivabradine — Ivabradine (5mg twice daily)
Drug: Conventional Treatment
  Arms: Group B Control Group

SUMMARY:
This study aims to evaluate the beneficial effect of heart rate reduction of oral ivabradine in patients presenting with non ST-segment elevation myocardial infarction (NSTEMI) during acute stage post percutaneous coronary intervention versus conventional treatment.

Materials and methods: A total of 100 patients admitted to the emergency department, National Heart Institute, Cairo, Egypt were randomized into two groups as follows: Group A: 50 patients with NSTEMI treated with ivabradine (5mg twice daily) in addition to the conventional treatment; Group B: 50 patients with NSTEMI treated with the conventional treatment only. Demographic data, detailed history, clinical examination, chest pain onset, blood pressure, heart rate (HR), temperature and respiratory rate, electrocardiogram (ECG) as well as echocardiography and laboratory investigations were recorded. Patients were monitored for a period of 3-5 days (acute stage).

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTEMI with normal sinus rhythm and heart rate (HR) more than 70 beats per minute (bpm) and systolic blood pressure (SBP) >90 mm Hg undergoing PCI

Exclusion Criteria:

* Patients needing urgent cardiac surgery, IV inotropic agents or had a HR less than 60 bpm without any medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate | acute stage post percutaneous coronary intervention (3-5 days)
  Heart Rate Reduction

IPD SHARING:
Plan to Share IPD: No